CLINICAL TRIAL: NCT03436238
Title: Myocardial Injury in Noncardiac Surgery in Sweden (MINSS) Study: Multi-centre, Observational Cohort Study of Patients Undergoing Elective, Major Abdominal Surgery.
Brief Title: Myocardial Injury in Noncardiac Surgery in Sweden
Acronym: MINSS
Status: Active, not recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other); Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Michelle Chew, Professor, Senior Consultant, Linkoeping University
Other Study IDs: MINSS
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Perioperative/Postoperative Complications; Risk Factor, Cardiovascular
Keywords: Perioperative; Biomarkers; Troponin; Prodrenomedullin; Endothelin; Perioperative Complications; Myocardial injury; Major adverse cardiovascular events
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MINSS cohort: Adult patients >= 50 years old undergoing elective, major, abdominal surgery requiring at least one overnight stay in hospital.
  Major abdominal surgery is defined as those classified as major OR major/complex by the Surgical Outcome Risk Tool (SORT) (www.sortsurgery.com).

SUMMARY:
The purpose of this multicentre, prospective, observational study is to identify robust biochemical markers that predict adverse cardiovascular outcomes and mortality in patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Inclusion Adults at least 50 years old undergoing elective, major or major/complex abdominal surgery defined according to the Surgical Outcome Risk Tool (www.sortsurgery.com), requiring general anaesthesia and at least one overnight stay. Exclusion Patients with acute coronary syndromes, new or decompensated heart failure at presentation, documented severeaortic stenosis, severely reduced ejection fraction (<40%) and inability to follow the procedures of the study or lack of capacity to give informed consent. Transplantation, trauma, endocrine, vascular and endovascular surgical procedures will also be excluded due to their distinct risk profiles compared with the intended population. Outcome The composite endpoint is all-cause mortality at 30 days and MACCE, the latter defined as nonfatal cardiac arrest, acute MI, congestive heart failure, new cardiac arrhythmia, angina and stroke. Secondary endpoints are 365-day all-cause mortality and MACCE. Data collection Relevant clinical and peri-operative data for example comorbidities, RCRI, ASA-PS score, type and length of surgery, blood loss and intra-operative lowest blood pressure will be collected.

Plasma levels of hsTnT, NTproBNP, Copeptin, MR-proADM and CT-proET1 will be measured at five sampling points: pre-operatively, immediately postoperatively, and on Days 1 to 3 postoperatively or until discharge. Data on MACCE will be obtained from patient records and structured telephone interviews at 30 and 365 days by assessors blinded to the results of the biomarker analyses.

Statistics Based on an assumed incidence of MINS of 10%(1) and 365-day mortality in the non-MINS group of 11% (estimate based on current data from the Swedish Perioperative Registry), the required sample size to detect an effect size of 10% is 1142. To account for drop-outs and missing data, we will recruit up to 1600 patients.

Receiver operating curve analysis will be used to determine the optimal threshold of each biomarker in predicting mortality/MACCE. The net reclassification index will be used to assess if biomarkers confer added value to the RCRI for the classification of MACCE.

A multivariable Cox proportional hazard models will be used to test the independent prognostic value of biomarkers. The sample size allows for adjustment of the following prespecified variables, selected on the basis of clinical plausibility and prior evidence: age, sex, ASA-PS class, RCRI, Charlson Comorbidity Index, length and type of surgery, presence of intra-operative hypotension, pre-operative creatinine and haemoglobin, biomarkers (alone and in combination). An independent statistical analysis will be conducted after recruitment of 600 patients to assess the frequency of outcomes and missing data, after which the sample size may be adjusted.

NOTE: An independent assessment by the Data Safety and Monitoring Board (DSMB) specifically addressing a revision of the sample size found that a total of 1269-1334 participants would be required for the study. This was based on a lower than expected rate of missing data (7.6% at DSMB assessment vs. expected 33% during study planning).

We therefore revised the sample size to 1269 (-1334) participants on 2 September 2019.

UPDATE 26 Feb 2022:

This study (including outcomes up to 30d after surgery) has been published: https://www.bjanaesthesia.org/article/S0007-0912(21)00649-8/fulltext

UPDATE 11 Jan 2023:

The following preplanned substudies are ongoing:

1. Effect of myocardial injury (MINS) on quality of recovery in patients undergoing major abdominal procedures in Sweden.

   The aim of the study is to investigate the postoperative quality of recovery (QoR) and the disability-free survival (DFS) among patients undergoing major abdominal surgery with and without perioperative myocardial injury in non-cardiac surgery (MINS). Our hypothesis is that patients with MINS have a poorer QoR and reduced DFS at short- and long-term follow-up.

   P:nested, cohort sub study within the Myocardial Injury in Noncardiac Surgery in Sweden (MINSS, NCT 03436238) study including patients from 2 participating hospitals E: Acute perioperative myocardial injury, defined as an increase in hsTnT≥14 ng L-1 above baseline value and measured at days 0-3 postoperatively.

   C: No perioperative myocardial injury O:Postoperative Quality of Recovery (QoR-15) scores at 7-10 days, 30-days and 1-year after surgery compared to the baseline. Secondary outcome is Disability Free Survival at 30-days and 1-year after surgery. DFS is defined as alive and WHODAS score of ≤ 25%.
2. The Effect of Perioperative Haemoglobin Decrease on Long-term Surgical Outcomes.

   The aim of this study is to investigate the effect of perioperative decrease in haemoglobin (Hb) level on the long-term outcomes of patients undergoing major abdominal surgery.

   P:We will include all patients enrolled in the MINSS study if there are available post-operative Hb measurement(s) and 1-year follow-up data.

   E:perioperative decrease in Hb level is the exposure variable of this study. C:various strata of perioperative Hb decrease O:The primary outcome of this study is the composite of one-year all-cause mortality and major adverse cardiovascular and cerebrovascular events (MACCE). The secondary outcome is 30-day post-operative complications defined as MACCE, re-operation, anastomosis leakage, post-operative infections or bleeding, renal or respiratory failure and pulmonary embolism
3. Incidence and trajectories of subclinical postoperative acute kidney injury (sPO-AKI), postoperative acute kidney injury (PO-AKI) and postoperative acute kidney disease (PO-AKD) among patients undergoing elective, major non-cardiac surgery.

   The primary aim of this study is to investigate the incidence of subclinical postoperative acute kidney injury (sPO-AKI), postoperative acute kidney injury (PO-AKI) and postoperative acute kidney disease (PO-AKD) and the trajectory of sPO-AKI, among patients undergoing elective, major non-cardiac surgery.

   Secondary aims are to evaluate the relationship between sPO-AKI and major adverse kidney events by 30 days (MAKE30) and all-cause mortality at 30 days postoperatively as well as chronic kidney disease (CKD) at one year postoperatively.

   P: nested, cohort sub study within the Myocardial Injury in Noncardiac Surgery in Sweden (MINSS, NCT 03436238) study including patients from 2 participating hospitals E:Serum creatinine (sCr) measured preoperatively and days 0-3 postoperatively, sCr obtained from patient charts between day 4-365 and occurrence of ICD codes N17.9, N18.X, N19.9 and N99.9 between day 0-365.

   C: no increase in sCr O: The primary outcome is incidence of sPO-AKI, PO-AKI and PO-AKD, as defined below.

   The secondary outcomes are 30-day all-cause mortality, MAKE 30, and CKD at 1-year post-surgery
4. The predictive role of MR-proADM for postoperative infections after major non-cardiac surgery: a sub-study of MINSS The primary aim of this study is to assess if mid-regional pro-adrenomedullin (MR-proADM) adds value to standard biomarkers in predicting postoperative infection following major non-cardiac surgery.

The secondary aim is to assess the prognostic value of MR-proADM for 30-day and 12-month all-cause mortality.

P:Predefined, nested sub-study of the Myocardial Injury in Noncardiac Surgery in Sweden project (MINSS, NCT 03436238) including patients from Linköping University and Norrköping Hospitals.

E: Increased plasma values of MR-proADM measured preoperatively and days 0-3 postoperatively.

C: No increase in plasma MR-proADM O:10-day postoperative infections Postoperative infections are defined as the presence of any of the following: superficial wound infections, deep wound infections, body cavity infections, pneumonias, urinary tract infections, bloodstream infections and sepsis as outlined in the European Perioperative Clinical Outcome (EPCO) 2014 definitions.

Secondary outcome:

30-day all-cause mortality. 12-month all-cause mortality. 10-day postoperative sepsis.

5) Phenotypes of perioperative myocardial injury and impact on long-term outcomes among patients undergoing major elective non-cardiac surgery.

The aim of this study is to evaluate how different phenotypes of myocardial injury may impact the long-term outcomes among patients undergoing major elective non-cardiac surgery. P: Pre-planned, sub-study within the Myocardial Injury in Noncardiac Surgery in Sweden (MINSS), a multicenter, prospective cohort study with available long-term follow-up data.

E:Patients are classified to 1) isolated preoperative increases (>99th URL) in hs-cTnT (likely chronic), 2) perioperative changes (postop-preop >99th URL) with normal preoperative hs-cTnT, 3) perioperative changes (postop-preop >99th URL) with increased preoperative hs-cTnT, 4) only postoperative increases (99th URL between 2 postoperative measurements.

C: no pre-, peri- or postoperative hs-cTnT increases O: The primary outcomes are all-cause mortality and major adverse cardiovascular and cerebrovascular events (MACCE) at longest follow up. MACCE is the composite of non-fatal cardiac arrest, myocardial infarction, new onset angina, new onset heart failure, new onset arrythmia (atrial fibrillation, atrial flutter, or second- or third-degree atrioventricular block), non-fatal cardiac arrest, and cerebrovascular insult (stroke and transient ischemic attack).

The secondary outcomes are the individual components of the MACCE definition described above, cardiac death (according to StEP COMPAC), and extracardiac adverse events (sepsis, acute kidney injury, pulmonary embolism) at longest follow up.

6) Incidence and outcome of perioperative blood transfusion in patients undergoing major non-cardiac surgery in Sweden. aims to investigate the incidence and outcome of perioperative blood transfusion in patients undergoing major non-cardiac surgery in Sweden. Proposed research questions will include:

1. What is the incidence of perioperative transfusion of blood and blood products?
2. What is the relationship between preoperative anaemia and intraoperative transfusion?
3. What is the relationship between preoperative anaemia and post-operative transfusion?
4. What is the relationship between intra- and post-operative transfusions and mortality, major adverse cardiovascular and cerebrovascular events and postoperative infections? P:nested cohort in the MINSS study including 3 participating centres E:perioperative blood transfusion C:no perioperative blood transfusion O:The primary outcome of this study is the transfusion of any blood product within the first 3 days of surgery. A co-primary outcome is the composite of all-cause mortality, major adverse cardiovascular and cerebrovascular events, and post-operative infection at 30 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective, major abdominal surgery*.

(*Major abdominal surgery requiring general anaesthesia, and requiring at least one overnight stay. Major abdominal surgery is defined as those classified as major OR major/complex by the Surgical Outcome Risk Tool (SORT) (www.sortsurgery.com).

In essence major surgery is one that penetrates and exposes a body cavity or produces a substantial impairment of physical or physiologic function or involves extensive dissection or transection. Examples of a major abdominal surgery include, but are not limited to, any procedure involving a laparotomy or laparoscopic procedures of the stomach, duodenum, small and large intestine and rectum. It also includes but is not limited to procedures on the reproductive system (total abdominal hysterectomy, salpingo-oophorectomy) and genitourinary system (nephrectomy, cystectomy).)

Exclusion Criteria:

* Patient not fulfilling inclusion study criteria above and/or clinician refusal and/or non-eligible as defined below.

Patients undergoing the following surgical procedures will NOT be eligible:

* transplantation
* trauma
* endocrine
* vascular
* endovascular

The presence of any one of the following will also lead to exclusion of the patient:

* ACS at presentation (clinical assessment or documentation)
* New or decompensated congestive heart failure at presentation (clinical assessment or documentation)
* Documented severe aortic stenosis (valve area < 1cm2)
* Reduced LVEF (<40%); if no LVEF is available, it will be assumed to be >40%
* Inability to follow the procedures of the study, e.g. due to language problems, dementia, etc. of the participant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective, major abdominal surgery at participating centres, requiring general anaesthesia, and requiring at least one overnight stay.
Sampling Method: Non-Probability Sample
Enrollment: 1269 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days post surgery
  All-cause mortality at 30 days post-surgery.
30-day MACCE | 30 days post surgery
  Major adverse cardio- cerebrovascular events (MACCE) at 30 days post-surgery.

SECONDARY OUTCOMES:
12-month mortality | 12 months post surgery
  All-cause mortality at 12 months post-surgery.
12-month MACCE | 12 months post surgery
  Major adverse cardio- cerebrovascular events (MACCE) at 12 months post-surgery.

OTHER OUTCOMES:
Net reclassification index (NRI) | 30 days post surgery
  The NRI will be calculated to assess if a preoperative elevated biomarker panel confers added value over RCRI
Long term mortality | 3 years and 5 years
  Long-term mortality will be extracted from the Swedish Registry of Deaths

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Chew, MBBS, PhD, Principal Investigator — Linkoeping University and Region Östergötland
Locations (7):
- Sweden (7):
  - Kristianstad KRYH Hospital, Kristianstad, Skåne County
  - Eskilstuna Hospital, Eskilstuna
  - Ryhov County Hospital, Jönköping
  - Skane University Hospital Lund, Lund
  - Skane University Hospital Malmö, Malmo
  - Vrinnevi Hospital, Norrköping
  - Department of Anaesthesia and Intensive Care, Linkoeping University Hospital, Region Östergötland, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Falt M, Ahman R, Hammarskjold F, Lyckner S, Jawad M, Andersson U, Fredrikson M, Sperber J, Elander L, De Geer L, Didriksson H, Jonsson C, Andersson H, Chew MS. Long-term outcomes of time-dependent phenotypes of perioperative myocardial injury☆. BJA Open. 2025 Jun 4;14:100422. doi: 10.1016/j.bjao.2025.100422. eCollection 2025 Jun. PMID 40529719
- [Derived] Chew MS, Puelacher C, Patel A, Hammarskjold F, Lyckner S, Kollind M, Jawad M, Andersson U, Fredrikson M, Sperber J, Johnsson P, Elander L, Zeuchner J, Linhardt M, De Geer L, Rolander WG, Gagno G, Didriksson H, Pearse R, Mueller C, Andersson H. Identification of myocardial injury using perioperative troponin surveillance in major noncardiac surgery and net benefit over the Revised Cardiac Risk Index. Br J Anaesth. 2022 Jan;128(1):26-36. doi: 10.1016/j.bja.2021.10.006. Epub 2021 Nov 29. PMID 34857357